CLINICAL TRIAL: NCT03986489
Title: Mindfulness-based Dance/Movement Therapy for Chronic Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Drexel University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Stony Brook University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1810006694; 7R34AT009555-02 (NIH)
Record Dates: First submitted 2019-05-29; First posted 2019-06-14 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2020-12

CONDITIONS: Chronic Low-back Pain
Keywords: Dance/movement therapy; Mindfulness-based dance/movement therapy; Chronic pain management; Creative Arts Therapies; Non-pharmacological intervention; Online intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based dance/movement therapy (Experimental): Participants assigned to the M-DMT group condition will receive care as usual plus 12 weekly 90-minute group M-DMT sessions delivered online by a board-certified dance/movement therapist. The therapist is instructed to follow the M-DMT manualized protocol.
  Interventions: Behavioral: Mindfulness-based dance/movement therapy (M-DMT)
- Chronic pain social support group (Active Comparator): Participants assigned to the control condition will participate in a 12-session (90-minute session/week) online social support group.
  Interventions: Behavioral: Chronic pain social support group

INTERVENTIONS:
Behavioral: Mindfulness-based dance/movement therapy (M-DMT) — M-DMT includes benefits of physical activity, group psychotherapy, mindfulness training, and an art-based intervention in a unified practice. Each online session focuses on different psycho-educational topics about chronic low back pain management and links these topics with specific M-DMT activities that incorporate mindfulness-based principles and techniques.
  Other Names: Dance/Movement Therapy
  Arms: Mindfulness-based dance/movement therapy
Behavioral: Chronic pain social support group — The therapist will facilitate online open group discussions about participants' experiences with or reactions to the topic of discussion and will promote empathy among group members. The therapist will use client-centered, reflective listening techniques but will not prescribe any specific recommendations for change.
  Each week, SSG participants will receive emails with brief information about the topic discussed during the group session.
  Arms: Chronic pain social support group

SUMMARY:
The purpose of this study is to evaluate the feasibility, acceptability and credibility of a mindfulness-based dance/movement therapy (M-DMT) protocol that is delivered online; to assess and improve methodological procedures for conducting a randomized controlled trial (RCT) test of M-DMT; and to demonstrate proof of principle by gathering information about the process of change between M-DMT and a control condition.

This is the first study to address the potential of M-DMT as a creative, non-opioid intervention for chronic back pain. Therefore, the findings of this study will provide important methodological and protocol data and substantive pilot data necessary for the next phase of this line of research, namely a fully powered RCT to evaluate efficacy and treatment mechanisms of action. Data obtained as part of this study will be instrumental for informing the systematic evaluation of M-DMT for chronic back pain care.

ELIGIBILITY:
Inclusion Criteria

* age > 18 years
* current non-specific cLBP that has persisted at least 3 months, and has resulted in pain on at least half the day in the past 6 months
* proficient in English
* average pain severity and interference ratings >3/10 on a 0-10 numeric rating scale
* if taking pain medication(s), dosage must be stabilized for a minimum of 3 months
* patients agree not to seek additional therapies for the duration of this study beyond those already included in their current treatment regimen or new treatments prescribed by their physician
* naïve to DMT.
* those who have adequate computer literacy (e.g., know how to use a computer to perform basic tasks such as open/send emails, use internet, fill-out online surveys) and access to the virtual delivery format (i.e., internet service and a personal computer device such as laptop, desktop, tablet PC).

Exclusion Criteria:

* pregnancy
* severe and/or progressive medical, neurological, substance dependence within the last 6 months or severe mental illness (i.e., psychosis, mania) that would prevent active participation
* cognitive impairment that prohibits informed consent
* back surgery in the last 6 months
* low back pain attributable to a recognizable, known specific pathology (e.g. infection, tumor, osteoporosis, fracture, structural deformity, inflammatory disorder, radicular syndrome, or cauda equina syndrome
* wheelchair-bound or unable to move without assistance
* involvement in impending litigation or judgment for disability or worker's compensation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Recruitment: Number of participants eligible | Baseline
  Number of participants eligible for randomization to the study intervention
Recruitment Rate | Baseline
  Proportion of participants randomized relative to total trial referrals
Recruitment time | Baseline
  Number of participate enrolled per month
Feasibility of recruiting male participants: Proportion of male participant enrolled | Baseline
  Proportion of male participant enrolled to the study
Treatment Completion Rate | 12 weeks following receipt of treatment
  We expect 80% of participants to complete at least 9/12 M-DMT sessions
Retention Rate | 24 weeks
  Proportion of participants who complete follow-up questionnaires
Reason for withdrawal | 12 weeks following receipt of treatment
  Assessed by an open-ended question, "What was the reason for discontinuing your participation?" administered by a study staff during a phone interview
M-DMT intervention credibility and expectancy | 1 week
  Credibility/Expectancy Questionnaire (range 3-27; higher scores reflect greater treatment expectancy and rationale credibility)
Treatment Fidelity | 1-12 weeks
  Treatment fidelity assessment form developed by the researcher (range: varies between sessions depending on the number of items included in the particular session; A total score of 80% and higher reflects adequate treatment fidelity)
Treatment satisfaction and acceptability: Likert-scale survey | 12 weeks post-randomization
  via Likert-scale surveys; on scale of 1 to 5, 1 being not satisfied; 5 being very satisfied (i.e higher number, better outcome).
M-DMT intervention acceptability | 12 weeks
  Exit interview based on an interview protocol developed by the researcher
Adverse Event | 1 -12 weeks
  Number of adverse events

SECONDARY OUTCOMES:
Pain intensity: PROMIS® Pain Intensity-Short Form (SF)3a | Change from Baseline pain intensity at 6, 12, and 24-week time points
  PROMIS® Pain Intensity-Short Form (SF)3a (A 5-point (from 1= Had no pain to 5= Very Severe) rating scale is used in each of the 3 items; higher results mean higher intensity of pain.
Pain interference: PROMIS® Pain Interference -8a | Change from Baseline pain interference at 6, 12, and 24-week time points
  PROMIS® Pain Interference -8a (A 5-point (from 1= Not at all to 5= Very much) rating scale is used on each of the 8 items; higher scores reflect greater pain interference
Chronic pain acceptance: Chronic Pain Acceptance Questionnaire | Change from Baseline chronic pain acceptance at 6, 12, and 24-week time points
  Chronic Pain Acceptance Questionnaire (A seven-point (from 0= Never to 6 = Always) rating scale is used in each of the 20 items; higher results mean high pain acceptance)
Mindfulness | Change from Baseline mindfulness at 6, 12, and 24-week time points
  Cognitive and Affective Mindfulness Scale (A 4-point (Rarely/not at all to almost always) rating scale is used in each of the 12 items; higher values reflect higher mindful qualities
Physical activity (Accelerometry data) | Change from Baseline physical activity at 12, and 24-week time points
  An accelerometer, ActiGraph GT9X will be used to measure the change in participants physical activity between baseline and 2 endpoints (12 and 24 weeks)
Physical activity (Self-report data) | Change from Baseline physical activity at 6, 12, and 24-week time points
  Self-report assessment of physical activity will be done through UCLA Activity Scale (One item out of 10 will be checked to best describe current activity level)

OTHER OUTCOMES:
Physical Function | Change from Baseline physical function at 6, 12, and 24-week time points
  PROMIS® Physical function-20a (A 5-point (5= without any difficulty to 1= Unable to do) rating scale is used in each of the 20 items; higher values reflect higher abilities to physically function
Depression | Change from Baseline depression at 6, 12, and 24-week time points
  PROMIS® Emotional Distress-Depression-SF 4a (A 5-point (1= Never to 5= Always) rating scale is used in each of the 4 items; higher values reflect higher levels of depression
Sleep Disturbance | Change from Baseline sleep disturbance at 6, 12, and 24-week time points
  PROMIS® Sleep Disturbance-4a (A 5-point (5= Very poor to 1= Very good) rating scale is used in each of the 4 items; higher values reflect higher levels of sleep disturbances
Pain Catastrophizing: Pain Catastrophizing Scale | Change from Baseline pain catastrophizing at 6, 12, and 24-week time points
  Pain Catastrophizing Scale - short form(SF)-4a (A 4-point (0= Not at all to 4= All the time) rating scale is used in each of the 4 items; higher scores reflect greater pain catastrophizing
Kinesiophobia | Change from Baseline kinesiophobia at 6, 12, and 24-week time points
  Tampa Scale of Kinesiophobia (A 4-point (1= Strongly disagree to 4= Strongly agree) rating scale is used in each of the 11 items; higher values reflect higher levels of kinesiophobia
Patient Perception of Change | 12 weeks
  Score on single item Patient Global Impression of Change Rating (range: 1 (No change) to 7 (a great deal better))

CONTACTS AND LOCATIONS:
Overall Officials: Minjung Shim, PhD, Principal Investigator — Drexel University; Adam Gonzalez, PhD, Principal Investigator — Stony Brook University
Locations (1):
- Drexel Universitsy, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No